CLINICAL TRIAL: NCT06745505
Title: EFFECTIVENESS of PRE-OPERATIVE BOWEL PREPARATION VS NO BOWEL PREPARATION on OUTCOMES of PEDIATRIC COLORECTAL SURGERIES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Collaborators: Holy Family Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Mansoor Ahmed, Resident Pediatric Surgery, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RMU-RRF-SUR002-23
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Surgery; Pediatric; Bowel Preparation
Keywords: effectiveness; pre-operative bowel preparation; pediatric colorectal surgery
MeSH Terms: interventions — Cathartics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Recieved Bowel Preparation (Experimental)
  Interventions: Procedure: Bowel Preparation
- Did not receive Bowel Preparation (Active Comparator)
  Interventions: Procedure: Bowel Preparation

INTERVENTIONS:
Procedure: Bowel Preparation — Group A received bowel preparation and Group B did not.

SUMMARY:
To compare the effectiveness of pre-operative bowel preparation vs no bowel preparation on outcomes of pediatric colorectal surgeries.

DETAILED DESCRIPTION:
Objective was to compare the effectiveness of pre-operative bowel preparation vs no bowel preparation on outcomes of pediatric colorectal surgeries. After approval from the ethical committee, 62 patients fulfilling the inclusion criteria were enrolled in this study from outpatient department. All participants were examined physically in person by the primary investigator. After which the patients were divided randomly into two groups A and B, 31 patients in each group. Group A patients were undergone bowel preparation while group B patients were not undergone bowel preparation. All patients were operated by a single consultant pediatric surgeon with more than 10 years of experience. Patients were called for follow up weekly till 6 weeks. Hospital stay was noted at the time of discharge. Wound infection rate was assessed till 30th post-operative day while anastomotic leak was ruled out on clinical and radiologic exam if symptoms were present. All the data of this study were analyzed in SPSS version 26. We concluded that that there is no significant difference in surgical outcomes between the group receiving the bowel preparation versus the group not receiving the bowel preparation in terms of surgical site infection rate, anastomotic leak and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients with congenital condition such as Hirschsprung disease, anorectal malformation requiring pull through with or without covering colostomy.
* Patients with anorectal malformation requiring anorectoplasty with or without covering colostomy.
* Ileostomy/colostomy acquired due to intestinal perforation, intestinal obstruction, and trauma admitted for reversal.
* Age up to 12 years.
* Patients of both genders.

Exclusion Criteria:

* Any associated congenital morbid anomaly having Meningomyelocoele, Muscular dystrophy (were assessed on clinical examination)
* Patients with behavior disorders such as autism (were assessed during psychiatric history and clinical examination)
* Patients with behavioral disorder are difficult to counsel and follow up

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
No difference in surgical outcome after bowel preparation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Salman Qamar, MBBS, Principal Investigator — Rawalpindi Medical College
Locations (1):
- Department of Pediatric Surgery, Holy Family Hospital, Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No